CLINICAL TRIAL: NCT00220779
Title: Randomized, Double-Blind, Placebo-Controlled Study to Compare the Effects of Different Dose Regimens of IGIV Chromatography (IGIV-C), 10% Treatment on Relapses in Patients With Relapsing Remitting Multiple Sclerosis
Brief Title: Immune Globulin Intravenous (IGIV) To Treat Relapsing, Remitting Multiple Sclerosis
Acronym: PRIVIG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 100434
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Results first posted 2014-04-11 (Estimated); Last update posted 2016-04-27 (Estimated); Status verified 2016-03

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — gamma-Globulins; Caprylates; Immunoglobulins, Intravenous; Immunoglobulins; Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1 (Experimental): IGIV-C 0.2 g/kg bw/infusion (2 ml/kg bw)
  Interventions: Drug: Immune Globulin IV [Human], 10% Caprylate/Chromatography Purified
- Group 2 (Experimental): IGIV-C 0.4 g/kg bw/infusion (4 ml/kg bw)
  Interventions: Drug: Immune Globulin IV [Human], 10% Caprylate/Chromatography Purified
- Group 3 (Placebo Comparator): placebo (0.1% albumin) 4 ml/kg bw/infusion
  Interventions: Drug: Albumin (Human) 25%, United States Pharmacopeia (USP)

INTERVENTIONS:
Drug: Immune Globulin IV [Human], 10% Caprylate/Chromatography Purified
  Other Names: Gamunex®; IGIVnex®; Gaminex; IGIV-C; Immune Globulin Intravenous (Human) , 10%; IGIV; BAY 41-1000; TAL-05-00004; IGIV-C, 10%; IVIG; Immune Globulin (Human), 10% (IGIV); Immune Globulin Intravenous, 10% by Chromatography Process; NDC 13533-645-12; NDC 13533-645-15; NDC 13533-645-20; NDC 13533-645-24; NDC 13533-645-71
  Arms: Group 1; Group 2
Drug: Albumin (Human) 25%, United States Pharmacopeia (USP)
  Other Names: Plasbumin®-5; Plasbumin®-25; Plasbumin®-5 (Low Aluminum); Plasbumin®-25 (Low Aluminum); Albumin (Human) 5%, USP; Albumin (Human) 25%, USP; TAL-05-00009; TAL-05-00023; TAL-05-00025; TAL-05-00026; BAY 34-9255; NDC 13533-684-16; NDC 13533-684-25; NDC 13533-684-71; NDC 13533-685-20; NDC 13533-685-25; NDC 13533-685-27; NDC 13533-690-20; NDC 13533-690-25; NDC 13533-690-27; NDC 13533-692-16; NDC 13533-692-20; NDC 13533-692-71
  Arms: Group 3

SUMMARY:
The trial will study 2 doses of Immune Globulin Intravenous (Human), 10% Caprylate/Chromatography Purified (IGIV-C) for the number of relapses that occur in a 1 year treatment period.

DETAILED DESCRIPTION:
This trial is designed as a multi-national, randomized, double-blind, placebo-controlled prospective trial with three parallel groups.

One hundred twenty (120) patients, 40 per treatment arm, with relapsing-remitting (RR) multiple sclerosis will be enrolled in this trial. Eligible patients must have a diagnosis of MS as per the McDonald Criteria. In addition, patients must have a diagnosis of relapsing-remitting course of MS defined as periods of worsening of neurological function with full recovery or with sequelae and residual deficit upon recovery; periods between disease relapses characterized by lack of disease progression. Patients must also have active disease with at least 1 defined documented relapse in the last year.

During a 2 month run-in period, 2 MRIs will be performed 6 weeks apart and patients will be stratified based on the presence or absence of 1 or more Gadolinium enhancing lesions on the first MRI (Gd-enhancing lesion yes-no) and will be randomized to one of two dose regimens of IGIV-C or matching placebo. Patients will receive study drug infusions every 4 weeks for 48 weeks for a total of 12 infusions. Patients will be evaluated by MRI every 6 weeks and by clinical assessments every 3 months. A follow-up visit will occur 4 weeks after the last infusion.

The treatment groups are as follows:

* IGIV-C - 0.2 g/kg body weight (bw)/infusion (2 ml/kg bw)
* IGIV-C - 0.4 g/kg bw/infusion (4 ml/kg bw)
* placebo (0.1% albumin) - 4 ml/kg bw/infusion

For blinding purposes, at each infusion, all patients will receive a total volume of 4 ml/kg bw. For patients receiving 0.2 g/kg bw of IGIV-C, the final volume of 4 ml/kg bw will be adjusted by the addition of dextrose 5%. Placebo will be supplied as Albumin 5% or Albumin 25% and diluted with either dextrose 5% or saline to a final concentration of 0.1% albumin.

Dose adaptation will be performed for subsequent infusions in case the patient's body weight has changed > 10%. The maximum amount available per infusion will be 400 ml (8 vials) calculated for a patient with a body weight of 100 kg. The suggested initial infusion rate will be 0.02 ml/kg/min for the first 15 minutes. If there is no evidence of a hypersensitivity reaction, the infusion may be given at a slowly increasing rate over the next 30 minutes up to a maximum allowable rate of 0.08 ml/kg/min. As such, the infusion for a 70 kg patient will take approximately 1hour 15 min. The overall infusion time may have a range from 1 to 2 hours.

ELIGIBILITY:
Inclusion Criteria:

* Symptoms consistent with Multiple Sclerosis up to 5 years
* Diagnosis of multiple sclerosis according to McDonald criteria.
* Diagnosis of relapsing-remitting (RR) multiple sclerosis (MS) (Defined as periods of worsening of neurological function with full recovery or with sequelae and residual deficit upon recovery; periods between disease relapses characterized by lack of disease progression
* Kurtzke Extended Disability Status Scale (EDSS) < 5.0
* At least 1 defined and documented relapse during the last year. Prior relapses where symptoms were due solely to a change in Bowel/Bladder Function or Cognitive Function will not be considered relapses as defined by this protocol and therefore not counted for inclusion into the study.
* Females or males; females of childbearing potential must use adequate contraception
* Clinically stable for at least 30 days prior to entry
* At least 9 hyperintense T2 lesions on MRI or 1 Gd-enhancing lesion according to McDonald/Barkhof dissemination-in-space criteria at entry
* Patients who have been informed about available treatments and decided, not to go on these treatments
* Written informed consent obtained prior to the initiation of any study related procedures

Exclusion Criteria:

* Females who are pregnant, breast feeding, or if, of childbearing potential, unwilling to practice adequate contraception throughout the study
* Prior therapy with azathioprine or any immunosuppressant agents within 6 months prior to study entry
* Prior steroid, methylprednisolone or adrenocorticotropic hormone (ACTH) therapy within 30 days prior to study entry
* Therapy with interferons (Betaseron®, Avonex®, Rebif®), glatiramer acetate (Copaxone®) or IGIV within 3 months prior to study entry or during the study
* Use of an investigational compound within 6 months prior to study entry
* Previous lymphoid irradiation or prior to treatment with cyclophosphamide, methotrexate or mitoxantrone
* Cardiac insufficiency (NYHA III/IV), cardiomyopathy, significant cardiac dysrhythmia requiring treatment, unstable or advanced ischemic heart disease (CCS III or IV), or malignant hypertension
* History of renal insufficiency or serum creatinine levels greater than 2.5 mg/dL (221 µmol/L)
* Known selective immunoglobulin A (IgA) deficiency or known antibodies to IgA
* Conditions whose symptoms and effects could alter protein catabolism and/or immunoglobulin G (IgG) utilization (e.g., protein-losing enteropathies, nephrotic syndrome)
* Any medical, psychiatric or other circumstances which impede or restrict the patient's participation in the study or any contraindication to contrast enhanced MRI (e.g.,pacemaker, aortic clip or any metal implant)
* Patients with clinically significant medical conditions including, but not limited to cardiac, pulmonary, hepatic, hematological (e.g. known coagulation disorder, history of deep venous thrombosis and/or pulmonary embolism), endocrine,or renal dysfunction, autoimmune disorders, severe environmental allergies or chronic infections

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 128 (Actual)
Dates: Start 2002-12; Primary Completion 2005-02 (Actual); Study Completion 2005-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fred D Lublin, MD, Principal Investigator — Mt Sinai Medical Center, New York, NY
Locations (37):
- United States (6):
  - Barrow Neurological Institute at St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Northwest NeuroSpecialists, PLLC, Tucson, Arizona
  - The Mt. Sinai Medical Center, Department of Neurology, New York, New York
  - SUNY Health Science Center at Stony Brook, Department of Neurology, Stony Brook, New York
  - Wake Forest University - School of Medicine, Winston-Salem, North Carolina
  - Neurology Health Care Service, Fletcher Allen Health Care, Burlington, Vermont
- Department of Neurology, Karl-Franzens University, Graz, Austria
- Canada (4):
  - Foothills Hospital, Calgary, Alberta
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, General Campus - Neurology Division, Ottawa, Ontario
  - CHUM Hospital Notre Dame, Montreal, Quebec
- Czechia (4):
  - Fakultni nemocnice Brno-Bohunice, Brno
  - St. Anna's Teaching Hospital, Brno
  - Všeobecná fakultní nemocnice, Prague
  - Department of Neurology, Motol Teaching Hospital, Prague
- Germany (7):
  - Medizinische Einrichtungen der Heinrich Heine Universitat, Neurologische Klinik, Düsseldorf
  - HELIOS Klinikum Erfurt GmbH, Klinik und Poliklinik fur Neurologie, Erfurt
  - Klinikum der Justus-Liebig-Universitat, Zentrum fur Neurologie und Neurochirurgie, Giessen
  - Universitatsklinikum Munster, Klinik und Poliklinik fur Neurologie, Münster
  - Klinikum Osnabrück GmbH, Osnabrück
  - Universitatsklinikum Ulm, Poliklinik fur Neurologie, Ulm
  - Klinijum der Universitat Wurzburg, Neurologische Klinik und Poliklinik, Würzburg
- Henry Dunant Hospital, Athens, Greece
- Hungary (4):
  - Szent Imre Korhaz Neurologia, Budapest
  - Uzsoki Street Hospital, Budapest
  - Jahn Ferenc Delpesti Teaching Hospital, Budapest
  - Szeged University of Science, Szeged
- Lady Davis Carmel Medical Center, Haifa, Israel
- Poland (4):
  - Katedra I Klinika Neurologii; Slaskiej Akademii Medycznej, Samodzielny Publiczny Centralny Szpital Kliniczny, Katowice-Ligota
  - Katedra I Klinika Neurologii, Univerytetu Medycznego w Lodzi, Lodz
  - Katedra I Klinika Neurologii, Lublin
  - Klinika Neurologiczna, Wojskowy Instut Medyczny, Warsaw
- Slovakia (2):
  - Fakultna menocnica Bratislava, Bratislava
  - Dererova nemocnica s Poliklinikou Nerologicka Klinika, Bratislava
- Sweden (2):
  - Lasarette Neurologiavdeling, Lund
  - Karilinska Sjukhuset, Stockholm
- University Hospital, Queens Medical Centre, Nottingham, United Kingdom

REFERENCES:
- [Result] Fazekas F, Lublin FD, Li D, Freedman MS, Hartung HP, Rieckmann P, Sorensen PS, Maas-Enriquez M, Sommerauer B, Hanna K; PRIVIG Study Group; UBC MS/MRI Research Group. Intravenous immunoglobulin in relapsing-remitting multiple sclerosis: a dose-finding trial. Neurology. 2008 Jul 22;71(4):265-71. doi: 10.1212/01.wnl.0000318281.98220.6f. PMID 18645164

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 31 study centers in Austria, Canada, Czech Republic, Germany, United Kingdom, Greece, Hungary, Israel, Poland, and the United States.
Groups:
- IGIV-C 0.2 g/kg bw/Infusion (2 mL/kg Body Weight); IGIV-C 0.4 g/kg bw/Infusion (4 mL/kg Body Weight); Placebo (0.1% Albumin) 4 mL/kg Body Weight/Infusion: Immune globulin (intravenous) (IGIV)
Period: Overall Study
Arm/Group | IGIV-C 0.2 g/kg bw/Infusion (2 mL/kg Body Weight) | IGIV-C 0.4 g/kg bw/Infusion (4 mL/kg Body Weight) | Placebo (0.1% Albumin) 4 mL/kg Body Weight/Infusion
Started | 45 | 42 | 41
Completed | 38 | 38 | 37
Not Completed | 7 | 4 | 4
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 4 | 1
Not completed — Non-compliance | 1 | 0 | 0
Not completed — Too time consuming | 1 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 2
Not completed — Lack of Efficacy | 3 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IGIV-C 0.2 g/kg bw/Infusion (2 mL/kg bw) | IGIV-C 0.4 g/kg bw/Infusion (4 mL/kg bw) | Placebo (0.1% Albumin) 4 mL/kg bw/Infusion | Total
Number analyzed (Participants) | 45 | 42 | 41 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 1 | 0 | 1
  Between 18 and 65 years | 45 | 41 | 41 | 127
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.9 (7.5) | 34.4 (7.9) | 33.0 (8.7) | 33.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 27 | 31 | 96
  Male | 7 | 15 | 10 | 32
Region of Enrollment [Number; unit: participants]
  United States | 5 | 3 | 3 | 11
  Czech Republic | 6 | 10 | 6 | 22
  Hungary | 4 | 2 | 2 | 8
  Greece | 1 | 2 | 0 | 3
  Canada | 5 | 1 | 5 | 11
  Poland | 10 | 6 | 8 | 24
  Austria | 3 | 1 | 2 | 6
  Israel | 1 | 0 | 2 | 3
  Germany | 9 | 15 | 11 | 35
  United Kingdom | 1 | 2 | 2 | 5

OUTCOME MEASURES:

1. Secondary Outcome: Effect on the Combined Unique Lesion Activity on Magnetic Resonance Imaging (MRI)
Time Frame: 1 year
Reporting Status: Not Posted

2. Primary Outcome: Percentage of Relapse Free Subjects (no Relapse)
Description: A relapse was defined for the purposes of this study as the appearance or reappearance of one or more neurological symptoms or worsening of an old symptom attributed to multiple sclerosis (MS) persisting for at least 48 hours and immediately preceded by a relatively stable or improving neurological state of at least 30 days.
Time Frame: 12 months
Population: Intent-to-Treat (ITT) Population was all randomized subjects. This was the primary analysis population.
Measure: Number; unit: percentage of participants
Arm/Group | IGIV-C 0.2 g/kg bw/Infusion (2 mL/kg bw) | IGIV-C 0.4 g/kg bw/Infusion (4 mL/kg bw) | Placebo (0.1% Albumin) 4 mL/kg bw/Infusion
Number analyzed (Participants) | 44 | 42 | 41
percentage of participants
  No Relapse | 56.8 | 59.5 | 68.3
  At Least One Relapse | 43.2 | 40.5 | 31.7
Statistical Analysis 1: Comparison: IGIV-C 0.2 g/kg bw/Infusion (2 mL/kg bw) vs Placebo (0.1% Albumin) 4 mL/kg bw/Infusion; The primary efficacy comparison was the comparison of the proportions of relapse free subjects (relapse defined as reported, not necessarily confirmed relapse). The multiple test procedure (hierarchical procedure) was to be stopped as soon as one of the statistical tests resulted in a non-significant P value > 0.05; Test type: Superiority or Other; p = 0.221, Cochran-Mantel-Haenszel — 0.2g/kg IGIV Group versus Placebo
Statistical Analysis 2: Comparison: IGIV-C 0.4 g/kg bw/Infusion (4 mL/kg bw) vs Placebo (0.1% Albumin) 4 mL/kg bw/Infusion; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.471, Cochran-Mantel-Haenszel — 0.4 g/kg IGIV Group versus Placebo

ADVERSE EVENTS:
Arm/Group | IGIV-C 0.2 g/kg bw/Infusion (2 mL/kg bw) | IGIV-C 0.4 g/kg bw/Infusion (4 mL/kg bw) | Placebo (0.1% Albumin) 4 mL/kg bw/Infusion
Serious Adverse Events (participants affected / at risk) | 2/45 | 2/42 | 1/41
Other Adverse Events (participants affected / at risk) | 32/45 | 26/42 | 29/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IGIV-C 0.2 g/kg bw/Infusion (2 mL/kg bw) (N=45) | IGIV-C 0.4 g/kg bw/Infusion (4 mL/kg bw) (N=42) | Placebo (0.1% Albumin) 4 mL/kg bw/Infusion (N=41)
Headache (General disorders) | 1 | 0 | 0 — Subject #2005
Herpes Zoster ophthalmic (Eye disorders) | 1 | 0 | 0 — Subject #506004
Vasculitis, peripheral (Vascular disorders) | 0 | 1 | 0 — Subject #502004
Panic attacks (Psychiatric disorders) | 0 | 1 | 0 — Subject #506003
Toothache (General disorders) | 0 | 0 | 1 — Subject #507003
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IGIV-C 0.2 g/kg bw/Infusion (2 mL/kg bw) (N=45) | IGIV-C 0.4 g/kg bw/Infusion (4 mL/kg bw) (N=42) | Placebo (0.1% Albumin) 4 mL/kg bw/Infusion (N=41)
Vertigo (Ear and labyrinth disorders) | 4 | 2 | 2
Nausea (Gastrointestinal disorders) | 2 | 5 | 0
Vomiting (Gastrointestinal disorders) | 1 | 4 | 0
Asthenia (General disorders) | 2 | 1 | 3
Fatigue (General disorders) | 5 | 2 | 5
Feeling cold (General disorders) | 4 | 1 | 0
Pyrexia (General disorders) | 3 | 3 | 0
Bronchitis (Infections and infestations) | 2 | 0 | 3
Influenza (Infections and infestations) | 2 | 1 | 5
Nasopharyngitis (Infections and infestations) | 9 | 7 | 11
Rhinitis (Infections and infestations) | 3 | 7 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 0 | 5
Urinary tract infection (Infections and infestations) | 1 | 6 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 2
Dizziness (Nervous system disorders) | 3 | 1 | 1
Headache (Nervous system disorders) | 7 | 5 | 6
Hypoaesthesia (Nervous system disorders) | 3 | 4 | 2
Paraesthesia (Nervous system disorders) | 4 | 1 | 4
Depression (Psychiatric disorders) | 1 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 4
Erythema (Skin and subcutaneous tissue disorders) | 0 | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator must send a draft manuscript of the publication or abstract to the sponsor thirty days in advance of submission in order to obtain approval prior to submission of the final version for publication. This will be reviewed promptly and approval will not be withheld unreasonably. In case of a difference of opinion between the sponsor and the investigator(s), the contents of the publication will be discussed in order to find a solution which satisfies both parties.